CLINICAL TRIAL: NCT01636986
Title: Impact of a Novel Silicone Hydrogel in Reducing Contact Lens-Related Dryness Symptoms in Existing Contact Lens Wearers
Brief Title: A Prospective Study of Two Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A00930
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-11

CONDITIONS: Myopia
Keywords: myopia; contact lenses; dry eyes; comfort; replacement
MeSH Terms: conditions — Myopia; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DT1 (Experimental): Delefilcon A contact lenses worn bilaterally on a daily wear, daily disposable basis for 4 weeks
  Interventions: Device: Delefilcon A contact lenses
- 1DAVM (Active Comparator): Etafilcon A contact lenses worn bilaterally on a daily wear, daily disposable basis for 4 weeks
  Interventions: Device: Etafilcon A contact lenses

INTERVENTIONS:
Device: Delefilcon A contact lenses — Silicone hydrogel contact lenses for daily wear, daily disposable use
  Other Names: DAILIES TOTAL1®
  Arms: DT1
Device: Etafilcon A contact lenses — Hydrogel contact lenses for daily wear, daily disposable use
  Other Names: 1-DAY ACUVUE® MOIST™
  Arms: 1DAVM

SUMMARY:
The purpose of this study was to evaluate the performance of a novel silicone hydrogel contact lens, DAILIES TOTAL1® (DT1) compared to the standard hydrogel material in 1-DAY ACUVUE® MOIST® (1DAVM) contact lens in contact lens wearers identified as having contact lens-related dryness symptoms.

DETAILED DESCRIPTION:
Three study visits occurred over the course of 28 ± 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age of consent and sign written Informed Consent Document and HIPAA form.
* Currently wearing soft contact lenses and identified as having contact lens-related dryness symptoms based upon responses to the Contact Lens Dry Eye Questionnaire.
* Wearing either daily disposable contact lenses or bi-weekly/monthly replacement contact lenses, daily wear use only (no extended wear use).
* Able to achieve distance visual acuity of at least 20/25 in each eye with study lenses in the available parameters, -0.50D to -6.00D.
* Willing to wear study lenses for at least 8 hours/day and at least 5 days/week.
* Willing and able to follow instructions and maintain the appointment schedule.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Neophyte or current wearer of DAILIES TOTAL1® or 1-DAY ACUVUE® MOIST™ contact lenses.
* Requires monovision or presbyopic correction.
* Any systemic or ocular disease or disorder complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study.
* Recent (within 7 days of enrollment) or current ocular infection, active ocular inflammation, glaucoma or preauricular lymphadenopathy.
* Clinically significant lash or lid abnormality.
* Systemic disease that, in the investigator's best judgment, would prohibit or confound safe contact lens wear.
* History of ocular surgery/trauma within the last 6 months.
* Topical or systemic antibiotics use within 7 days of enrollment.
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kern, Ph.D., Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 US study center.
Pre-assignment Details: This reporting group includes all enrolled and randomized participants.
Groups:
- DAILIES TOTAL1: Delefilcon A contact lenses worn bilaterally on a daily wear, daily disposable basis for 4 weeks
Period: Overall Study
Arm/Group | DAILIES TOTAL1 | 1DAVM
Started | 30 | 32
Completed | 30 | 30
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Corneal Staining | 0 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled and randomized participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | DAILIES TOTAL1 | 1DAVM | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.26 (4.28) | 24.53 (4.83) | 23.89 (4.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Subjective Contact Lens-related Dryness Symptoms at Week 4 as Assessed by the CLDEQ
Description: Contact lens symptoms were evaluated using the Contact Lens and Dry Eye Questionnaire (CLDEQ). The participant indicated the frequency with which 9 common contact lens-related ocular surface dryness symptoms were experienced over the previous week. Each symptom was rated on a 5-point scale (1=never, 5=constantly). Both eyes contributed to the mean. A more negative change number indicates a greater perceived improvement, namely, lessening of the symptom.
Time Frame: Day 0, Week 4
Population: All enrolled and randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DAILIES TOTAL1 | 1DAVM
Number analyzed (Participants) | 30 | 30
Units on a scale
  Eyes feel uncomfortable | -0.21 (0.13) | -0.17 (0.16)
  Eyes feel dry | -1.07 (0.68) | -0.92 (0.90)
  Vision change between clear and blurry | -0.04 (0.04) | -0.04 (0.04)
  Eyes feel irritated | -0.42 (0.32) | -0.31 (0.28)
  Eyes feel gritty and scratchy | -0.10 (0.10) | -0.07 (0.07)
  Feel "something" in the eye | -0.47 (0.58) | -0.38 (0.54)
  Eyes burning and stinging | -0.25 (0.34) | -0.28 (0.36)
  Eyes feel unusually sensitive to bright light | -0.23 (0.35) | -0.19 (0.32)
  Eyes itch | -0.43 (0.41) | -0.38 (0.46)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (4 months).
Description: This reporting group includes all enrolled participants who were exposed to the test product.
Arm/Group | DAILIES TOTAL1 | 1DAVM
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 7/30 | 8/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DAILIES TOTAL1 (N=30) | 1DAVM (N=32)
Contact lens fell out (Eye disorders) | 0 | 2
Eye irritation (Eye disorders) | 4 | 4
Corneal Staining (Eye disorders) | 1 | 2
Foreign body sensation (Eye disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was not powered to detect differences in individual items.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.